CLINICAL TRIAL: NCT01351909
Title: Phase I Trial of Low-Dose Cyclophosphamide in Combination With Veliparib (ABT-888) in HER2/Neu-Negative Metastatic Breast Cancer
Brief Title: Cyclophosphamide and Veliparib in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02590; NCI-2011-02590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P8853_A18PAMDREVW01; 11-02-068; 11-01501; CDR0000700033; 8853 (Other: Montefiore Medical Center - Moses Campus); 8853 (Other: CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Unresectable Breast Carcinoma; Metastatic Breast Carcinoma; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (veliparib, cyclophosphamide) (Experimental): Patients receive veliparib orally PO QD and cyclophosphamide PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Veliparib

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of cyclophosphamide and veliparib when given together in treating patients with breast cancer that has spread from where it started to nearby tissue or lymph nodes or to other places in the body. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cyclophosphamide together with veliparib may work better in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of veliparib (ABT-888) that can be combined with metronomic dose cyclophosphamide in patients with metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To determine whether the macroH2A1.1 and poly (adenosine diphosphate [ADP]-ribose) polymerase 1 (PARP1) expression status in archival paraffin embedded tumor specimens from either the primary tumor or metastatic disease is predictive of clinical benefit with veliparib (ABT-888) plus cyclophosphamide.

OUTLINE: This is a dose-escalation study.

Patients receive veliparib orally (PO) once daily (QD) and cyclophosphamide PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Patients must have histologically confirmed breast cancer (metastatic breast cancer [MBC]) that is human epidermal growth factor receptor 2 (HER2/neu) negative (as determined by local pathology or reference laboratory), and have disease that is metastatic (stage IV [TxNxM1]) or locally advanced and not amenable to potentially curative surgical resection (eg, clinical stage IIIB-C)
* HER2/neu negative disease (performed on primary tumor and/or metastatic lesion using commercially available/approved assay in local institutional or reference laboratory), according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* National Comprehensive Cancer Network (NCCN) guidelines recommend for metastatic breast cancer "…biopsy documentation of first recurrence, if possible, and determination of hormone receptor status (estrogen receptor [ER] and progesterone receptor [PR]) and HER2 status…."; therefore, histologic and/or cytologic confirmation of metastatic disease is encouraged whenever feasible, but not required; in some circumstances, histologic confirmation may not be feasible (eg, bone metastases not amenable to biopsy and elevated cancer antigen [CA]27-29 tumor marker); for patients who have had histologic confirmation of metastatic disease, it is required that the biopsy confirm that the metastatic tumor is ER and/or PR positive, and HER2/neu negative; for patients in whom biopsy confirmation of metastatic disease is not feasible, it is required that the primary tumor be ER and/or PR-positive and HER2/neu negative
* Measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) or non-measurable disease, with measurement obtained within 4 weeks of registration
* Phase I: Patients must have received at least one prior chemotherapy regimen for metastatic disease; patients with deleterious germ line mutations in breast cancer (BRCA)1 or BRCA2 are not required to have received prior chemotherapy for metastatic disease
* Patients must have had progressive disease after at least one line of endocrine therapy for metastatic disease (includes relapse while receiving endocrine therapy); there should be at least 1 week interval between the last endocrine treatment for an aromatase inhibitor and at least 2 weeks for tamoxifen or fulvestrant
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dl (per manufacturer recommendation)
* Total bilirubin within normal institutional limits (unless isolated indirect hyperbilirubinemia due to Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients with a history of brain metastases are eligible if they have been treated with radiation and have stable brain metastases at least 3 months after radiation and must also be off steroids
* Patients must be able to swallow whole capsules and tolerate oral medications
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; being not of childbearing potential is defined as: (1) prior hysterectomy, or (2) no menstrual period for at least 24 months; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have radiotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to systemic agents administered more than 3 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases with active symptoms or requiring anticonvulsive medications, or steroids should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib (ABT-888) or cyclophosphamide used in the study
* Evidence of complete or partial bowel obstruction or other unable to take oral medications
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* Patients unable to swallow whole capsules
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant (positive pregnancy test) or lactating women will be excluded from the study; also, unwillingness to use effective means of contraception in subjects with child-bearing potential will be excluded from the study; women of child-bearing potential must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation
* Patients with active severe infection; known infection with human immunodeficiency virus (HIV), hepatitis B virus, hepatitis C virus, or severe concurrent illness will be excluded from the study; HIV-positive patients on combination antiretroviral therapy are ineligible
* Patients with a history of seizure disorder requiring antiepileptics who have had a seizure episode within the last 6 months
* Prior treatment with veliparib (ABT-888) or other PARP inhibitors (e.g., olaparib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of veliparib and cyclophosphamide | 21 days
  The descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 will be utilized for adverse events reporting.

SECONDARY OUTCOMES:
Clinical response (complete or partial response) according to RECIST version 1.1 | Up to 24 weeks
  Clinical response and benefit rates in each group will be estimated by computing proportions and corresponding 95% confidence intervals. Rates will be compared between groups using the Fisher's exact test.
Overall survival | Time from treatment initiation to death, assessed up to 6 years
  Overall survival will be analyzed using standard survival analytic approaches including the Kaplan-Meier method and the log-rank test.
MacroH2A1.1 expression levels | Up to 6 years
  Expression levels of macroH2A1.1 will be compared between patients with and without clinical benefit using the two-sample T-test or Wilcoxon rank sum test, depending on the distribution of the data. Logistic regression models will also be fit to the data to adjust for potential confounders in the analysis.
PARP1 expression status | Up to 6 years
  Expression levels of PARP1 will be compared between patients with and without clinical benefit using the two-sample T-test or Wilcoxon rank sum test, depending on the distribution of the data. Logistic regression models will also be fit to the data to adjust for potential confounders in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Sparano, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (5):
- United States (5):
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York